CLINICAL TRIAL: NCT06342882
Title: Functional Independence Levels Associated With Dysphagia Severity in Patients With Neurological Diseases
Brief Title: Dysphagia Severity and Functional Independence Level
Status: Completed | Type: Observational
Sponsor: Atılım University (Other)
Responsible Party: Sponsor
Other Study IDs: GO 19/833- A
Record Dates: First submitted 2024-02-19; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Dysphagia; Neurologic Disorder
Keywords: dysphagia; functional independance
MeSH Terms: conditions — Deglutition Disorders; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with dysphagia (study): In this study, patients who received PAS score 1 were included in the group without dysphagia (control group); and patients who were scored between 2 to 8 were included in the group with dysphagia (study group).
  Interventions: Diagnostic Test: dysphagia assessment; Diagnostic Test: functional independence level
- patients without dysphagia (control): In this study, patients who received PAS score 1 were included in the group without dysphagia (control group); and patients who were scored between 2 to 8 were included in the group with dysphagia (study group).
  Interventions: Diagnostic Test: dysphagia assessment; Diagnostic Test: functional independence level

INTERVENTIONS:
Diagnostic Test: dysphagia assessment — Twenty-one patients underwent the Modified Barium Swallowing Study and Swallowing Ability and Function Evaluation (SAFE) assessments. The Penetration Aspiration Scale (PAS) and SAFE physical examination, oral phase and pharyngeal phase domains was used to determine the dysphagia severity.
Diagnostic Test: functional independence level — Functional independence was evaluated by the Functional Independence Measurement (FIM) motor and cognitive domains.

SUMMARY:
Functional independence is the ability of a person to perform daily life activities safely without any restriction, as much as possible. The functional independence depends on physical, social, cognitive and psychological abilities of the person. Therefore, full functional independence requires the harmony of all these parameters.

Dysphagia can be seen in more than 50% of neurological patients, and it is called neurogenic dysphagia. Muscle weakness, tonus changes, sensory loss and coordination problems occur in these patients. Pain and fatigue are also frequently observe. These patients have problems with fine and gross motor movements, and thereby mobility and transfer activities become difficult. Life-threatening complications such as pulmonary problems, malnutrition and dehydration accompany when patients have dysphagia. Both neurological and dysphagia-related problems negatively affect the physical, psychological, emotional and cognitive functions of patients. Neurological patients with dysphagia may have more serious clinical situations due to more affected vital functions such as pulmonary functions and feeding.

Dysphagia-induced malnutrition adversely affects many systems, including the musculoskeletal system. In a study conducted in the elderly with dysphagia, atrophy in the total muscle mass and swallowing muscles, and increase in intramuscular adipose tissue were reported as a result of malnutrition. Decreases in the muscle mass may negatively affect the functional independence of patients with dysphagia. Other studies in geriatric population have shown that swallowing function is associated with hand grip strength and quadriceps muscle strength, which are indicators of functional independence in activities of daily living (ADL). These studies also suggest that dysphagia may be associated with functional independence in geriatric group. Therefore, functional independence may also reduce in patients with neurogenic dysphagia. However, there is no study investigating the relationship between dysphagia severity and the functional independence levels in patients with neurological diseases. Therefore, the investigators aimed to investigate the relationship between dysphagia severity and functional independence level in patients with neurological diseases.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18-65 years
* independent to walk 3 meters
* underwent a Modified Barium Swallowing Study (MBSS).

Exclusion Criteria:

* having any cervical pathology that may affect swallowing physiology,
* history of rheumatological diseases
* having any orthopedic surgery in the previous 6 months
* using a wheelchair.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neurological disorders
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
dysphagia severity | 1 day
  Swallowing Study and Swallowing Ability and Function Evaluation (SAFE) assessments. The SAFE physical examination, oral phase and pharyngeal phase domains was used to determine the dysphagia severity.
functional independence | 1 day
  Functional independence was evaluated by the Functional Independence Measurement (FIM) motor and cognitive domains.

CONTACTS AND LOCATIONS:
Overall Officials: selen serel arslan, Prof, Study Director — Hacettepe University
Locations (1):
- Atılım Uiveristy, Ankara, Incek, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided